CLINICAL TRIAL: NCT05350488
Title: Qualitative Analysis of the Post-Stroke Continuum Among African Stroke Survivors in Alabama
Status: Withdrawn | Type: Observational
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Danny Lee, Clinical Research Administrator II, University of Alabama at Birmingham
Other Study IDs: 300009035
Record Dates: First submitted 2022-03-30; First posted 2022-04-28 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Stroke; Disability Physical; Patient Satisfaction; Caregiver Burden
Keywords: Rehabilitation; Post-Stroke Rehabilitation Continuum
MeSH Terms: conditions — Stroke; Patient Satisfaction; Caregiver Burden | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stroke Survivors <1 year: Group A will include participants that are less than 1 year out from their most recent stroke.
  Interventions: Other: Informational Interview
- Stroke Survivors >1 year: Group B will include participants that are greater than 1 year out from their most recent
  Interventions: Other: Informational Interview
- Caregivers: Group C will include participants' identified caregivers.
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Informational Interview — Interview topics will fall in the broad categories of assessing medical knowledge and understanding of stroke, knowledge of medical and community resources, understanding and experience of post-stroke rehabilitation barriers faced upon reintegrating back home and ability to continue management of stroke diagnosis and suggestions for improvement.
  Groups: Stroke Survivors <1 year; Stroke Survivors >1 year
Other: Focus Group — Focus group topics will fall into the same broad categories as the informational interviews, however will be asked from a caregiver's perspective
  Groups: Caregivers

SUMMARY:
This proposal seeks to improve the investigators' post-stroke TOC process through developing an innovative, patient informed and guided solution aimed at addressing the investigators' deep south African American population within the UAB system. The investigators will engage participants in both urban and rural Alabama through informational interviews and work to find common themes to address so that future interventions are useful to their unique needs and desires. This goes beyond simply identifying barriers and endeavors to discovering solutions.

ELIGIBILITY:
Inclusion Criteria:

1. African American
2. Aged 40 years and older
3. Required home health therapy, outpatient therapy, skilled nursing facility or inpatient rehabilitation
4. Alabama Resident
5. Fluent in English
6. Stroke confirmed by advanced imaging (CT, MRI)
7. Zoom capability (participants can either have video conference ability or can call into Zoom line)
8. Caregivers must be identified by patients as providing a significant portion of care and/or be able to articulate their role as a caregiver

Exclusion Criteria:

1. Did not require home health therapy, outpatient therapy or inpatient rehabilitation
2. Long term residents of skilled nursing facility
3. Severe aphasia
4. Severe cognitive impairments

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will screen 60-100 individuals with the goal of enrolling a total of 20 AA stroke survivors +/- their identified caregivers. Individuals will be recruited from within the UAB Health System from the acute care neurology stroke service and the PI's stroke recovery clinic. Participants will be separated into 3 groups. Group A will include n=10 participants that are less than 1 year out from their most recent stroke. Group B will include n=10 participants that are greater than 1 year out from their most recent stroke. Group C will include the participants' identified caregivers. Having an available caregiver is preferred but is not required. Therefore, a goal of at least 10 caregivers is set.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment and retention | July 1,2022-January 20, 2023
  The investigators will screen 60-100 individuals with the goal of enrolling a total of 20 AA (African American) stroke survivors +/- their identified caregivers. Historically, there has been low recruitment and retention rates for AAs. The investigators plan to over-recruit in order to account for this phenomenon and track our success/failure rates with percent retained vs recruited.
Ability to use Zoom platform | July 1,2022-January 20, 2023
  The Zoom platform is becoming a more popular avenue to conduct qualitative interviews for research purposes among researchers and participants. The investigators will evaluate if this reported phenomenon is reproducible within this particular research cohort. Success will measured by a 50% or greater completion of interview and the ability to successfully connect to the zoom platform either via smart device or telephone dial in. The investigators will also document any technical difficulties that are encountered from either the interviewer's standpoint or the participant's standpoint.
Validity of questions asked to arrive at the themes that will appropriately inform the basis of this proposal | February 2023-May 2023
  We will extract data from transcriptions of participants' Zoom interviews and perform thematic analysis